CLINICAL TRIAL: NCT00199940
Title: A Pilot Open Trial Of Ziprasidone, Early In The Course Of Pediatric Psychotic Illness
Brief Title: Safety And Efficacy Study Of Ziprasidone In Pediatric Psychotic Illness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHW 03/162, HRRC 538-03
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2008-03-12 (Estimated); Status verified 2008-03

CONDITIONS: Schizophrenia; Affective Disorders; Psychotic Disorder; Psychotic Mood Disorder
Keywords: Schizophrenia; Pediatric psychotic disorders; Ziprasidone
MeSH Terms: conditions — Schizophrenia; Mood Disorders; Psychotic Disorders; Affective Disorders, Psychotic | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ziprasidone

SUMMARY:
The purpose of this research is to determine if Ziprasidone is safe and effective for use in children and adolescents with a psychotic illness, and to determine of Ziprasidone treatment leads to weight changes in children.

DETAILED DESCRIPTION:
Ziprasidone is a recently FDA approved antipsychotic, and it holds promise in the treatment of pediatric psychosis due to its low liability for weight gain and other side effects. This is important because early intervention in persons with a psychotic illness is important for their long-term treatment and outcome. Unfortunately, pediatric samples are often more sensitive to the side effects of psychotropic medications. Because psychotropic medications are often used by clinicians long before they are studied in pediatric populations, it is important to further study these agents.

Twenty subjects with the diagnosis of a psychotic disorder, according to DSM-IV criteria, will be recruited for the study. If subjects have completed baseline evaluations, labs, EKG, and rating scales and are still eligible to participate, subjects will start on 20mg of Ziprasidone at night. The second week this will increase to 20 mg twice a day. At visits that occur at 2,4,6,and 8 weeks, the subject's dose of medication can be increased in 20mg per day increments. This allows for a maximum possible dose of 100mg. Dosage may be decreased at any time secondary to side effects.

The potential benefits are that new information will be added to the field of pediatric psychiatry and the possibility that the medication may result in improved symptoms of psychosis. The potential benefits of this study outweigh the possible risks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia, Schizophreniform DO, Schizoaffective DO or Psychotic Disorder NOS
* Male/female, ages 7.0-17 years old
* Normal intelligence, ability to provide assent and consent
* Not currently receiving adequate treatment

Exclusion Criteria:

* Known hypersensitivity to ziprasidone (past failed trial)
* History of QTc prolongation
* Recent myocardial infarction
* Uncompensated heart failure
* Currently treated with other QTc prolonging medications
* Unstable medical illness
* If on diuretics, monitor regularly for hypokalemia

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 2003-12; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Symptom Scale (PANSS), score symptoms from baseline through end of study Week 8.

SECONDARY OUTCOMES:
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS), assess at baseline only.
Child Depression Rating Scale (CDRS), rate from baseline to Week 8.
Simpson-Angus Rating Scale (SARS), rate from baseline to Week 8.
Abnormal Involuntary Movement Scale (AIMS), rate at baseline, Weeks 2,4,6,8.
Barnes Akathesia Scale (BAS), rate from baseline through Week 8.
Side-Effect For Children & Adolescents (SEFCA), rate from baseline through Week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Russell E Scheffer, MD, Principal Investigator — Medical College of Wisconsin; Children's Hospital of Wisconsin